CLINICAL TRIAL: NCT03258294
Title: Effect of Melatonin on Sleep Disturbances in Patients With Parkinson's Disease: Double Blind, Randomized, Placebo Controlled Trial
Brief Title: Effect of Melatonin on Sleep Disturbances in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KIMJisun (Other)
Collaborators: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, KIMJisun, Instructor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-09-098-010
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
Keywords: melatonin; sleep disturbances
MeSH Terms: conditions — Parkinson Disease; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin(Circadin®) (Experimental): Melatonin(Circadin®) is taken orally, once daily before going to sleep for a period of 4 weeks.
  Interventions: Drug: Melatonin(Circadin®)
- Placebo (Placebo Comparator): Placebo tablet is taken orally, once daily before going to sleep for a period of 4 weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Melatonin(Circadin®)
  Arms: Melatonin(Circadin®)
Drug: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
This clinical study is a double-blind, randomized, placebo-controlled trial to investigate the effects of melatonin on the sleep disturbance symptoms of Parkinson's disease patients, symptoms which have a significant impact on the quality of life of these patients.

DETAILED DESCRIPTION:
After selecting patients who satisfied the inclusion criteria and were not disqualified by the exclusion criteria, through a double-blind procedure the patients are directed to orally take either the investigational drug melatonin or a placebo(allocation ratio 1:1) for 4 weeks, once daily, before going to sleep. The evaluation of efficacy and safety is performed at the first baseline and immediately after administering the drug for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the clinical criteria for idiopathic Parkinson's disease (United Kingdom Parkinson's Disease Brain Bank Criteria)
2. Patients who complain of sleep disturbances such as insomnia, REM sleep behavior disorder, excessive daytime sleepiness (EDS), etc.
3. Patients who have received drug treatment for at least 6 months since their diagnosis
4. Male or female patient aged 55 or older
5. Patients who have given voluntary consent after understanding the content of the clinical trial (in the case of elderly patients aged 70 or older, consent must be received from both the subject and the his or her legal representative)

Exclusion Criteria:

1. Patients with a serious cognitive disorder, behavioral disorder, or mental illness
2. Patients with a serious medical disease

   * Patients who concomitantly suffer from severe renal impairment, convulsions, stomach ulcers, moderate or more severe liver disease
   * Patients with un-controlled high blood pressure or diabetes
3. Patients who have taken another investigational products within 4 weeks prior to being enrolled in this clinical trial, or patients who are pregnant or breastfeeding
4. Patients who have a history of hypersensitivity to the investigational products or a drug similar in component or who have had heavy metal poisoning

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2016-01-13 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Variation in PSQI(Pittsburgh Sleep Quality Index) | Baseline and immediately after administering the drug for 4 weeks
  Variation in PSQI before and immediately after the administration of the drug

SECONDARY OUTCOMES:
Variations in RBDQ(The REM sleep Behavior Disorder screening Questionnaire) | Baseline and immediately after administering the drug for 4 weeks
Variations in PDSS(The Parkinson's Disease Sleep Scale) | Baseline and immediately after administering the drug for 4 weeks
Variations in ESS(The Epworth Sleepiness Scale) | Baseline and immediately after administering the drug for 4 weeks
Variations in UPDRS(Unified Parkinson Disease Rating Scale) | Baseline and immediately after administering the drug for 4 weeks
Variations in H & Y Scale(Hoehn and Yahr Scale) | Baseline and immediately after administering the drug for 4 weeks
Variations in NMSS(Non-Motor Symptom assessment Scale) | Baseline and immediately after administering the drug for 4 weeks
Variations in PDQ-39(The 39-Item Parkinson's Disease Questionnaire) | Baseline and immediately after administering the drug for 4 weeks

OTHER OUTCOMES:
Variations in CGI(Clinical Global Impression) | Baseline and immediately after administering the drug for 4 weeks
Variations in PGI(Patient Global Impression) | Baseline and immediately after administering the drug for 4 weeks
Number of subjects with adverse events | 4 weeks of drug treatment
Number of subjects with serious adverse events | 4 weeks of drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jisun Kim, Principal Investigator — Samsung Medical Center, Department of Neurology; Eungseok Oh, Principal Investigator — Chungnam National University Hospital, Department of Neurology; Wooyoung Jang, Principal Investigator — Gangneung Asan Hospital, Department of Neurology; Jinse Park, Principal Investigator — Inje University Haeundae Paik Hospital, Department of Neurology

IPD SHARING:
Plan to Share IPD: No